CLINICAL TRIAL: NCT00398034
Title: Analgesic Efficacy of Testosterone Replacement in Hypogonadal Opioid-treated Chronic Pain Patients: A Pilot Study.
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The original PI (David Siegel) Left the VA
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Solvay Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Chris Cardozo, Staff Physician, James J. Peters Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2192-06-049
Record Dates: First submitted 2006-11-08; First posted 2006-11-10 (Estimated); Last update posted 2023-10-13 (Actual); Status verified 2006-11

CONDITIONS: Pain; Hypogonadism
Keywords: opioids; pain; hypogonadism; depression; fatigue; cognition; libido
MeSH Terms: conditions — Pain; Hypogonadism; Depression; Fatigue

INTERVENTIONS:
Drug: Testosterone Gel

SUMMARY:
The purpose of this pilot study is to test the effects of testosterone replacement on pain, fatigue, mood, cognition and libido in hypogonadal men on long-term opioid therapy for chronic pain.

DETAILED DESCRIPTION:
Opioids are increasingly used for the treatment of non-malignant chronic pain with as many as five to ten million patients treated at the time of the most recent estimate in 2002. The side effects of opioids such as fatigue, loss of libido, Impaired cognition and sexual dysfunction have long been recognize and strikingly, resemble symptoms of hypogonadism in men. Many studies have demonstrated a high prevalence of hypogonadism in male subjects who are long-term users of opioids. The aims of this pilot study are, in hypogonadal men being treated with opioids for chronic pain, to: 1) determine the effect of TRT on pain; 2) determine effects of TRT on fatigue; 3) determine the effect of TRT on mood; 4) determine effects of TRT on cognition and 5) characterize the effects of TRT on sexual dysfunction. This study is a randomized, placebo-controlled, 6-week pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Adult male patients (above 18 years old and below 60 years old)
* Receiving greater than 20 IV morphine equivalents/day with <20% change in dosage in the last month.
* AM total testosterone <300 ng/dL
* Report "worst pain during the past week" grater than 4 on an 11-point numeric scale.

Exclusion Criteria:

* Females
* Poorly controlled, symptomatic, active medical or psychiatric problems (e.g., HIV, hepatitis, diabetes, cancer, benign prostatic hypertrophy, substance abuse, major depression)
* Neurological or psychiatric disorder that would compromise the patient's ability to give informed consent or adhere to the requirements of the protocol.
* History of prostate cancer, abnormal findings on digital rectal exam, or PSA greater than 4.0 ng/m
* History of polycythemia
* Renal or hepatic dysfunction
* Hematocrit >55%
* Known history of hypersensitivity to transdermal testosterone gel.
* Abnormalities during digital rectal exam.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2006-10-30 (Actual); Primary Completion 2007-09-06 (Actual); Study Completion 2007-09-06 (Actual)

PRIMARY OUTCOMES:
• To determine if testosterone replacement can improve pain control in opioid-treated, hypogonadal men with chronic pain.

SECONDARY OUTCOMES:
In opioid-treated, hypogonadal men with chronic pain, to determine whether testosterone replacement therapy (TRT) will:
reduce the opioid requirement.
improve fatigue
improve depression
improve sexual function.
Improve cognition
To determine the proportion of responders to the analgesic effects of TRT

CONTACTS AND LOCATIONS:
Overall Officials: Christopher P Cardozo, M.D., Principal Investigator — James J. Peters VAMC

REFERENCES:
- [Background] American Pain Society, Guidelines for the Management of Acute and Cancer Pain. 4 ed. 1999, Glenview, IL: American Pain Society.
- [Background] Portenoy RK. Opioid therapy for chronic nonmalignant pain: a review of the critical issues. J Pain Symptom Manage. 1996 Apr;11(4):203-17. doi: 10.1016/0885-3924(95)00187-5. PMID 8869456
- [Background] Rigoni, G. Drug Utilization for Immediate- and Modified Release Opioids in the U.S. in FDA Anesthesia, Life Support, and Addiction Drug Products Advisory Committee. 2003. Gaithersburg, Maryland.
- [Background] Bair MJ, Robinson RL, Katon W, Kroenke K. Depression and pain comorbidity: a literature review. Arch Intern Med. 2003 Nov 10;163(20):2433-45. doi: 10.1001/archinte.163.20.2433. PMID 14609780
- [Background] Passchier J, Rupreht J, Koenders ME, Olree M, Luitwieler RL, Bonke B. Patient-controlled analgesia (PCA) leads to more postoperative pain relief, but also to more fatigue and less vigour. Acta Anaesthesiol Scand. 1993 Oct;37(7):659-63. doi: 10.1111/j.1399-6576.1993.tb03784.x. PMID 8249554
- [Background] Jarvik LF, Simpson JH, Guthrie D, Liston EH. Morphine, experimental pain, and psychological reactions. Psychopharmacology (Berl). 1981;75(2):124-31. doi: 10.1007/BF00432173. PMID 6798601
- [Background] Cicero TJ, Bell RD, Wiest WG, Allison JH, Polakoski K, Robins E. Function of the male sex organs in heroin and methadone users. N Engl J Med. 1975 Apr 24;292(17):882-7. doi: 10.1056/NEJM197504242921703. PMID 1117911
- [Background] Crowley TJ, Simpson R. Methadone dose and human sexual behavior. Int J Addict. 1978 Feb;13(2):285-95. doi: 10.3109/10826087809039281. PMID 640760
- [Background] Cushman P Jr. Sexual behavior in heroin addiction and methadone maintenance. Correlation with plasma luteinizing hormone. N Y State J Med. 1972 Jun 1;72(11):1261-5. No abstract available. PMID 4503902
- [Background] Mintz J, O'Hare K, O'Brien CP, Goldschmidt J. Sexual problems of heroin addicts. Arch Gen Psychiatry. 1974 Nov;31(5):700-3. doi: 10.1001/archpsyc.1974.01760170088014. No abstract available. PMID 4474860
- [Background] Smith DE, Moser C, Wesson DR, Apter M, Buxton ME, Davison JV, Orgel M, Buffum J. A clinical guide to the diagnosis and treatment of heroin-related sexual dysfunction. J Psychoactive Drugs. 1982 Jan-Jun;14(1-2):91-9. doi: 10.1080/02791072.1982.10471916. PMID 7119946
- [Background] Azizi F, Vagenakis AG, Longcope C, Ingbar SH, Braverman LE. Decreased serum testosterone concentration in male heroin and methadone addicts. Steroids. 1973 Oct;22(4):467-72. doi: 10.1016/0039-128x(73)90002-0. No abstract available. PMID 4747447
- [Background] Bolelli G, Lafisca S, Flamigni C, Lodi S, Franceschetti F, Filicori M, Mosca R. Heroin addiction: relationship between the plasma levels of testosterone, dihydrotestosterone, androstenedione, LH, FSH, and the plasma concentration of heroin. Toxicology. 1979 Dec;15(1):19-29. doi: 10.1016/0300-483x(79)90016-7. PMID 120622
- [Background] Cushman P Jr. Plasma testosterone in narcotic addiction. Am J Med. 1973 Oct;55(3):452-8. doi: 10.1016/0002-9343(73)90202-7. No abstract available. PMID 4743346
- [Background] Mendelson JH, Mendelson JE, Patch VD. Plasma testosterone levels in heroin addiction and during methadone maintenance. J Pharmacol Exp Ther. 1975 Jan;192(1):211-17. PMID 1123724
- [Background] Rasheed A, Tareen IA. Effects of heroin on thyroid function, cortisol and testosterone level in addicts. Pol J Pharmacol. 1995 Sep-Oct;47(5):441-4. PMID 8868137
- [Background] Afrasiabi MA, Flomm M, Friedlander H, Valenta LJ. Endocrine studies in heroin addicts. Psychoneuroendocrinology. 1979;4(2):145-53. doi: 10.1016/0306-4530(79)90028-3. No abstract available. PMID 230529
- [Background] Brambilla F, Sacchetti E, Brunetta M. Pituitary-gonadal function in heroin addicts. Neuropsychobiology. 1977;3(2-3):160-6. doi: 10.1159/000117601. PMID 331136
- [Background] Mendelson JH, Mello NK. Plasma testosterone levels during chronic heroin use and protracted abstinence: study of Hong Kong addicts. NIDA Res Monogr. 1978;(19):142-8. No abstract available. PMID 106283
- [Background] Ragni G, De Lauretis L, Bestetti O, Sghedoni D, Gambaro V. Gonadal function in male heroin and methadone addicts. Int J Androl. 1988 Apr;11(2):93-100. doi: 10.1111/j.1365-2605.1988.tb00984.x. PMID 3372047
- [Background] Cushman P Jr, Kreek MJ. Methadone-maintained patients. Effect of methadone on plasma testosterone, FSH, LH, and prolactin. N Y State J Med. 1974 Oct;74(11):1970-3. PMID 4528642
- [Background] Daniell HW. Narcotic-induced hypogonadism during therapy for heroin addiction. J Addict Dis. 2002;21(4):47-53. doi: 10.1300/J069v21n04_05. PMID 12296501
- [Background] Lafisca S, Bolelli G, Franceschetti F, Filicori M, Flamigni C, Marigo M. Hormone levels in methadone-treated drug addicts. Drug Alcohol Depend. 1981 Nov;8(3):229-34. doi: 10.1016/0376-8716(81)90066-1. PMID 6459917
- [Background] Kley HK, Oellerich M, Wiegelmann W, Herrmann J, Rudorff KH, Nieschlag E, Kruskemper HL. The effect of methadone on hypophyseal and peripheral glandular hormones during withdrawal. Horm Metab Res. 1977 Nov;9(6):484-8. doi: 10.1055/s-0028-1093505. No abstract available. PMID 412765
- [Background] Woody G, McLellan AT, O'Brien C, Persky H, Stevens G, Arndt I, Carroff S. Hormone secretion in methadone-dependent and abstinent patients. NIDA Res Monogr. 1988;81:216-23. No abstract available. PMID 3136363
- [Background] Daniell HW. Hypogonadism in men consuming sustained-action oral opioids. J Pain. 2002 Oct;3(5):377-84. doi: 10.1054/jpai.2002.126790. PMID 14622741
- [Background] Rajagopal A, Vassilopoulou-Sellin R, Palmer JL, Kaur G, Bruera E. Hypogonadism and sexual dysfunction in male cancer survivors receiving chronic opioid therapy. J Pain Symptom Manage. 2003 Nov;26(5):1055-61. doi: 10.1016/s0885-3924(03)00331-2. PMID 14585556
- [Background] Abs R, Verhelst J, Maeyaert J, Van Buyten JP, Opsomer F, Adriaensen H, Verlooy J, Van Havenbergh T, Smet M, Van Acker K. Endocrine consequences of long-term intrathecal administration of opioids. J Clin Endocrinol Metab. 2000 Jun;85(6):2215-22. doi: 10.1210/jcem.85.6.6615. PMID 10852454
- [Background] Finch PM, Roberts LJ, Price L, Hadlow NC, Pullan PT. Hypogonadism in patients treated with intrathecal morphine. Clin J Pain. 2000 Sep;16(3):251-4. doi: 10.1097/00002508-200009000-00011. PMID 11014399
- [Background] Paice JA, Penn RD, Ryan WG. Altered sexual function and decreased testosterone in patients receiving intraspinal opioids. J Pain Symptom Manage. 1994 Feb;9(2):126-31. doi: 10.1016/0885-3924(94)90166-x. PMID 7517429
- [Background] Roberts LJ, Finch PM, Pullan PT, Bhagat CI, Price LM. Sex hormone suppression by intrathecal opioids: a prospective study. Clin J Pain. 2002 May-Jun;18(3):144-8. doi: 10.1097/00002508-200205000-00002. PMID 12048415
- [Background] Mendelson JH, Inturrisi CE, Renault P, Senay EC. Effects of acetylmethadol on plasma testosterone. Clin Pharmacol Ther. 1976 Mar;19(3):371-4. doi: 10.1002/cpt1976193371. PMID 1261171
- [Background] Mendelson JH, Ellingboe J, Judson BA, Goldstein A. Plasma testosterone and luteinizing hormone levels during levo-alpha-acetylmethadol maintenance and withdrawal. Clin Pharmacol Ther. 1984 Apr;35(4):545-7. doi: 10.1038/clpt.1984.75. PMID 6705455
- [Background] Yilmaz B, Konar V, Kutlu S, Sandal S, Canpolat S, Gezen MR, Kelestimur H. Influence of chronic morphine exposure on serum LH, FSH, testosterone levels, and body and testicular weights in the developing male rat. Arch Androl. 1999 Nov-Dec;43(3):189-96. doi: 10.1080/014850199262481. PMID 10624501
- [Background] Adams ML, Sewing B, Forman JB, Meyer ER, Cicero TJ. Opioid-induced suppression of rat testicular function. J Pharmacol Exp Ther. 1993 Jul;266(1):323-8. PMID 8392556
- [Background] Khan C, Malik SA, Iqbal MA. Testosterone suppression by heroin. J Pak Med Assoc. 1990 Jul;40(7):172-3. No abstract available. PMID 2125664
- [Background] Malik SA, Khan C, Jabbar A, Iqbal A. Heroin addiction and sex hormones in males. J Pak Med Assoc. 1992 Sep;42(9):210-2. PMID 1433805
- [Background] Cicero TJ, Wilcox CE, Bell RD, Meyer ER. Acute reductions in serum testosterone levels by narcotics in the male rat: stereospecificity, blockade by naloxone and tolerance. J Pharmacol Exp Ther. 1976 Aug;198(2):340-6. PMID 948030
- [Background] Cicero TJ, Badger TM. A comparative analysis of the effects of narcotics, alcohol and the barbiturates on the hypothalamic-pituitary-gonadal axis. Adv Exp Med Biol. 1977;85B:95-115. doi: 10.1007/978-1-4615-9038-5_8. PMID 596294
- [Background] Cicero TJ, Meyer ER, Wiest WG, Olney JW, Bell RD. Effects of chronic morphine administration on the reproductive system of the male rat. J Pharmacol Exp Ther. 1975 Mar;192(3):542-8. PMID 1168254
- [Background] Cicero TJ, Bell RD, Meyer ER, Schweitzer J. Narcotics and the hypothalamic-pituitary-gonadal axix: acute effects on luteinizing hormone, testosterone and androgen-dependent systems. J Pharmacol Exp Ther. 1977 Apr;201(1):76-83. PMID 850146
- [Background] Cicero TJ, Badger TM, Wilcox CE, Bell RD, Meyer ER. Morphine decreases luteinizing hormone by an action on the hypothalamic-pituitary axis. J Pharmacol Exp Ther. 1977 Dec;203(3):548-55. No abstract available. PMID 336869
- [Background] Murphy MR. Methadone reduces sexual performances and sexual motivation in the male Syrian golden hamster. Pharmacol Biochem Behav. 1981 Apr;14(4):561-7. doi: 10.1016/0091-3057(81)90317-8. PMID 7232476
- [Background] Mendelson JH, Ellingboe J, Kuehnle J, Mello NK. Heroin and naltrexone effects on pituitary-gonadal hormones in man: tolerance and supersensitivity. NIDA Res Monogr. 1979;27:302-8. No abstract available. PMID 121347
- [Background] Mendelson JH, Ellingboe J, Keuhnle JC, Mello NK. Effects of naltrexone on mood and neuroendocrine function in normal adult males. Psychoneuroendocrinology. 1978 Oct;3(3-4):231-6. doi: 10.1016/0306-4530(78)90013-6. No abstract available. PMID 219434
- [Background] Catlin DH, Poland RE, Gorelick DA, Gerner RH, Hui KK, Rubin RT, Li CH. Intravenous infusion of beta-endorphin increases serum prolactin, but not growth hormone or cortisol, in depressed subjects and withdrawing methadone addicts. J Clin Endocrinol Metab. 1980 Jun;50(6):1021-5. doi: 10.1210/jcem-50-6-1021. PMID 7372783
- [Background] Grossman A. Brain opiates and neuroendocrine function. Clin Endocrinol Metab. 1983 Nov;12(3):725-46. doi: 10.1016/s0300-595x(83)80062-0. PMID 6323067
- [Background] Mendelson JH, Meyer RE, Ellingboe J, Mirin SM, McDougle M. Effects of heroin and methadone on plasma cortisol and testosterone. J Pharmacol Exp Ther. 1975 Nov;195(2):296-302. PMID 1185598
- [Background] Mirin SM, Meyer RE, Mendelson JH, Ellingboe J. Opiate use and sexual function. Am J Psychiatry. 1980 Aug;137(8):909-15. doi: 10.1176/ajp.137.8.909. PMID 6774622
- [Background] Morley JE. The endocrinology of the opiates and opioid peptides. Metabolism. 1981 Feb;30(2):195-209. doi: 10.1016/0026-0495(81)90172-4. PMID 6258010
- [Background] Oyama T, Toyota M, Shinozaki Y, Kudo T. Effects of morphine and ketamine anaesthesia and surgery on plasma concentrations of luteinizing hormone, testosterone and cortisol in man. Br J Anaesth. 1977 Oct;49(10):983-90. doi: 10.1093/bja/49.10.983. PMID 921876
- [Background] Su CF, Liu MY, Lin MT. Intraventricular morphine produces pain relief, hypothermia, hyperglycaemia and increased prolactin and growth hormone levels in patients with cancer pain. J Neurol. 1987 Dec;235(2):105-8. doi: 10.1007/BF00718020. PMID 3430186
- [Background] von Graffenried B, del Pozo E, Roubicek J, Krebs E, Poldinger W, Burmeister P, Kerp L. Effects of the synthetic enkephalin analogue FK 33-824 in man. Nature. 1978 Apr 20;272(5655):729-30. doi: 10.1038/272729a0. No abstract available. PMID 643067
- [Background] Cicero TJ. Effects of exogenous and endogenous opiates on the hypothalamic--pituitary--gonadal axis in the male. Fed Proc. 1980 Jun;39(8):2551-4. PMID 6247215
- [Background] Purohit V, Singh HH, Ahluwalia BS. Failure of methadone-treated human testes to respond to the stimulatory effect of human chorionic gonadotrophin on testosterone biosynthesis in vitro. J Endocrinol. 1978 Aug;78(2):299-300. doi: 10.1677/joe.0.0780299. No abstract available. PMID 702024
- [Background] Ragni G, De Lauretis L, Gambaro V, Di Pietro R, Bestetti O, Recalcati F, Papetti C. Semen evaluation in heroin and methadone addicts. Acta Eur Fertil. 1985 Jul-Aug;16(4):245-9. PMID 4072581
- [Background] Couzinet B, Schaison G. The control of gonadotrophin secretion by ovarian steroids. Hum Reprod. 1993 Nov;8 Suppl 2:97-101. doi: 10.1093/humrep/8.suppl_2.97. PMID 8276977
- [Background] Martini L, Motta M, Piva F, Zanisi M. LHRF, LHRH, GnRH: what controls the secretion of this hormone? Mol Psychiatry. 1997 Sep;2(5):373-6. doi: 10.1038/sj.mp.4000311. PMID 9322226
- [Background] Yen SS, Quigley ME, Reid RL, Ropert JF, Cetel NS. Neuroendocrinology of opioid peptides and their role in the control of gonadotropin and prolactin secretion. Am J Obstet Gynecol. 1985 Jun 15;152(4):485-93. doi: 10.1016/s0002-9378(85)80162-9. PMID 2990210
- [Background] Rasmussen DD, Liu JH, Wolf PL, Yen SS. Endogenous opioid regulation of gonadotropin-releasing hormone release from the human fetal hypothalamus in vitro. J Clin Endocrinol Metab. 1983 Nov;57(5):881-4. doi: 10.1210/jcem-57-5-881. PMID 6311863
- [Background] Ebeling PR. Osteoporosis in men. New insights into aetiology, pathogenesis, prevention and management. Drugs Aging. 1998 Dec;13(6):421-34. doi: 10.2165/00002512-199813060-00002. PMID 9883398
- [Background] Anderson FH. Osteoporosis in men. Int J Clin Pract. 1998 Apr-May;52(3):176-80. PMID 9684434
- [Background] Elhassan AM, Lindgren JU, Hultenby K, Bergstrom J, Adem A. Methionine-enkephalin in bone and joint tissues. J Bone Miner Res. 1998 Jan;13(1):88-95. doi: 10.1359/jbmr.1998.13.1.88. PMID 9443794
- [Background] Perez-Castrillon JL, Olmos JM, Gomez JJ, Barrallo A, Riancho JA, Perera L, Valero C, Amado JA, Gonzalez-Macias J. Expression of opioid receptors in osteoblast-like MG-63 cells, and effects of different opioid agonists on alkaline phosphatase and osteocalcin secretion by these cells. Neuroendocrinology. 2000 Sep;72(3):187-94. doi: 10.1159/000054586. PMID 11025413
- [Background] Rico H, Costales C, Cabranes JA, Escudero M. Lower serum osteocalcin levels in pregnant drug users and their newborns at the time of delivery. Obstet Gynecol. 1990 Jun;75(6):998-1000. PMID 2342747
- [Background] Pedrazzoni M, Vescovi PP, Maninetti L, Michelini M, Zaniboni G, Pioli G, Costi D, Alfano FS, Passeri M. Effects of chronic heroin abuse on bone and mineral metabolism. Acta Endocrinol (Copenh). 1993 Jul;129(1):42-5. doi: 10.1530/acta.0.1290042. PMID 8351958
- [Background] Miller K, Corcoran C, Armstrong C, Caramelli K, Anderson E, Cotton D, Basgoz N, Hirschhorn L, Tuomala R, Schoenfeld D, Daugherty C, Mazer N, Grinspoon S. Transdermal testosterone administration in women with acquired immunodeficiency syndrome wasting: a pilot study. J Clin Endocrinol Metab. 1998 Aug;83(8):2717-25. doi: 10.1210/jcem.83.8.5051. PMID 9709937
- [Background] Forman LJ, Tingle V, Estilow S, Cater J. The response to analgesia testing is affected by gonadal steroids in the rat. Life Sci. 1989;45(5):447-54. doi: 10.1016/0024-3205(89)90631-0. PMID 2770410
- [Background] Frye CA, Seliga AM. Testosterone increases analgesia, anxiolysis, and cognitive performance of male rats. Cogn Affect Behav Neurosci. 2001 Dec;1(4):371-81. doi: 10.3758/cabn.1.4.371. PMID 12467088
- [Background] Stoffel EC, Ulibarri CM, Craft RM. Gonadal steroid hormone modulation of nociception, morphine antinociception and reproductive indices in male and female rats. Pain. 2003 Jun;103(3):285-302. doi: 10.1016/s0304-3959(02)00457-8. PMID 12791435